CLINICAL TRIAL: NCT07235280
Title: An Open-Label Safety and Tolerability Pilot Study of Dapagliflozin in Stage IA Lung Adenocarcinoma
Brief Title: Testing the Safety of Dapagliflozin Prior to Surgery for the Treatment of Patients With Stage IA Lung Adenocarcinoma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-1048; NCI-2025-07570 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Lung Adenocarcinoma; Stage IA1 Lung Cancer American Joint Committee on Cancer (AJCC) v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Lung Neoplasms | interventions — Specimen Handling; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (dapagliflozin) (Experimental): Patients receive dapagliflozin PO QD for 30 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT-guided biopsy on study and collection of blood and urine samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography Assisted Biopsy; Drug: Dapagliflozin Propanediol; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and urine samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography Assisted Biopsy — Undergo CT-guided biopsy
  Other Names: Computed Tomography Biopsy; Computed Tomography-Guided Needle Biopsy; CT Assisted Biopsy; CT Guided Biopsy
Drug: Dapagliflozin Propanediol — Given PO
  Other Names: Dapagliflozin Propylene Glycol Hydrate; Dapagliflozin S-propylene Glycol Monohydrate; Farxiga
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This early phase I trial tests the safety and side effects of dapagliflozin given prior to surgery in patients with stage IA lung adenocarcinoma. Dapagliflozin is approved by the Food and Drug Administration (FDA) for the treatment of diabetes and heart failure. It is an SGLT2 inhibitor. Stage I lung adenocarcinomas express significantly higher levels of the SGLT2 protein than other stages, and research suggests that SGLT2 inhibition improves lung cancer outcomes in patients with diabetes. In this study, dapagliflozin is being used off-label, which means it is being used for a condition that it was not originally approved for by the FDA. The investigational study drug is a neoadjuvant treatment, meaning the drug is given before surgery to try and help make the surgery more effective.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess safety and tolerability of administering 30 days of neoadjuvant dapagliflozin propanediol (dapagliflozin) before surgery in subjects with stage Ia lung adenocarcinoma.

SECONDARY OBJECTIVE:

I. To measure the effects of dapagliflozin on tumor cell proliferation in lung adenocarcinoma.

EXPLORATORY OBJECTIVES:

I. To measure the effects of neoadjuvant dapagliflozin on biological and metabolic parameters.

II. To measure the effects of neoadjuvant dapagliflozin on biomarkers.

OUTLINE:

Patients receive dapagliflozin orally (PO) once daily (QD) for 30 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT)-guided biopsy on study and collection of blood and urine samples throughout the study.

After completion of study treatment, patients are followed up between days 64 and 72.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide written informed consent
* Male or female ≥ 22 years of age at visit 1
* Histologically confirmed stage Ia lung adenocarcinoma, with availability of biopsy tissue for Ki-67 determination
* Planning to undergo surgery for lung adenocarcinoma
* Willing and able to receive a research CT-guided lung biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Leukocytes ≥ 3.0 K/mm^3
* Absolute neutrophil count ≥ 1.5 K/mm^3
* Platelets ≥ 100 K/mm^3
* Total bilirubin ≤ 2 mg/dl
* Aspartate aminotransferase (AST) ≤ 62 IU/L
* Alanine aminotransferase (ALT) ≤ 70 IU/L
* Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73m^2
* Diabetic status: diabetic subjects who are not currently receiving treatment will be included in the study. Diabetic subjects who are under treatment with insulin or oral anti-diabetic drugs will be enrolled under observation by endocrinologists on the team, to adjust the dose of the standard of care diabetic drugs to prevent hypoglycemia
* Females of child-bearing potential must have a negative pregnancy test during screening and be neither breastfeeding nor intending to become pregnant during study participation. Females of childbearing potential must agree to avoid pregnancy during the study and omit to abstinence from heterosexual intercourse or agree to use two methods of birth control (one highly effective method and one additional effective method) at least 4 weeks before the start of protocol therapy
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study. Women of child-bearing age will receive a urine pregnancy test to confirm eligibility
* Unsuitable candidate for the study, based on the opinion of the Investigator (e.g., cognitive impairment), such that participation might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements or complete the study
* Current or previous treatment with SGLT2 inhibitors
* History of other malignancies with exception of malignancies for which all treatment was completed at least 2 years before registration with no evidence of disease and locally treated skin squamous or basal cell carcinoma
* Currently receiving any other investigational agents
* Currently receiving regularly scheduled systemic steroids in the form of prednisone or dexamethasone (more than 10 mg prednisone daily or equivalent). Topical steroid ointments or creams for occasional skin rash is allowed
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to dapagliflozin
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, ketoacidosis, severe kidney disease (estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73m^2)
* Subjects with HIV are eligible unless their cluster of differentiation 4 (CD4+) T-cell counts are < 350 cells/µL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective antiretroviral therapy (ART) according to Department of Health and Human Services (DHHS) treatment guidelines is recommended

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to day 64-72
  Will be measured by frequency and severity of toxicities related to dapagliflozin per Common Terminology Criteria for Adverse Events version 6.0. Data will be summarized. Adverse events, severe adverse events, and adverse drug reactions will be coded by body system and Medical Dictionary for Regulatory Activities classification term. Adverse events will be tabulated and will include the number of patients for whom the event occurred, the rate of occurrence, and the severity and relationship to study drug.

SECONDARY OUTCOMES:
Tumor cell proliferation change | From biopsy to surgery up to day 64-72
  Tumor cell proliferation change will be measured by percentage of Ki-67-positive cells at 3 separate timepoints: 1. pre-treatment archival tissue of standard of care diagnostic lung biopsy samples; 2. pre-treatment research computed tomography-guided lung biopsy; 3. post-treatment archival tissue from the standard of care lung tissue sample from the surgical resection. Will utilize mixed effect negative binomial regression models to compare the Ki-67 in pre- versus post-investigational study drug treatment lung biopsy samples. The outcome in these models will be the number of Ki-67 positive cells in the lung biopsy. The primary inference for the efficacy of the treatment will be the time effect in the model which will test whether the rate of Ki-67 positivity changes is due to the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Scafoglio, MD/PhD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center; Jane Yanagawa, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States